CLINICAL TRIAL: NCT04588207
Title: Urea for Chronic Hyponatremia: A Pilot Study
Brief Title: Urea for Chronic Hyponatremia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to recruit participants
Sponsor: Helbert Rondon Berrios, MD, MS (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Helbert Rondon Berrios, MD, MS, Associate Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20050035; R21DK122023 (NIH)
Record Dates: First submitted 2020-10-07; First posted 2020-10-19 (Actual); Results first posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-04

CONDITIONS: Hyponatremia; Inappropriate ADH Syndrome
Keywords: Hyponatremia; SIADH; SIAD; Urea
MeSH Terms: conditions — Hyponatremia; Inappropriate ADH Syndrome | interventions — Urea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- On Urea, Then Off Urea (Experimental): Participants assigned to this group will receive oral urea for 42 days (period 1), followed by a 10-day washout period, and then will be off urea for 42 days (period 2).
  Interventions: Drug: Urea
- Off Urea, Then On Urea (Experimental): Participants assigned to this group will be off urea during for 42 days (period 1), followed by a 10-day washout period, and then on urea for 42 days (period 2)
  Interventions: Drug: Urea

INTERVENTIONS:
Drug: Urea — Groups "On Urea, Then Off Urea" and "Off Urea, Then On Urea" will receive urea during period 1 and period 2 of the study, respectively. The investigators will use the new American formulation of oral urea (i.e., Ure-Na™), which is packaged as a powder and mixed with 4 ounces. of water for oral consumption. Urea will be started at a dose of 15 grams of urea per mouth once daily. Dose titration will be based on the absolute increase in PNa on days 7 and 14. The urea dosing scheme will involve increasing from the starting dose of 15 grams/day to 30 grams/day (in 2 divided doses) based on the change in and absolute value of PNa, and subsequently, from 30 grams/day to 60 grams/day (in 2 divided doses) when indicated. The maximal dose of urea administered will be 60 g/day.
  Other Names: Ure-Na

SUMMARY:
This study is examining how a dietary supplement called urea can be used to treat low blood sodium level. Low blood sodium level is a common problem and some studies show that many patients with low blood sodium level suffer from brain fog and/or loss of balance. Unfortunately, it is unknown at this point what the best treatment is for low blood sodium level. With this pilot research study, the investigators are hoping to learn more about whether urea is safe to take, whether patients can tolerate taking urea for several weeks, whether urea increases blood sodium level, and whether urea can help prevent the brain fog and/or loss of balance that some patients with low blood sodium level suffer from. The information obtained with this study is intended to be used to design a larger study in the future to get a definite answer whether urea is beneficial for patients with low blood sodium level.

DETAILED DESCRIPTION:
Hyponatremia is the most common electrolyte disorder encountered clinically. While acute and/or severe hyponatremia is commonly associated with significant symptoms, milder and more chronic forms of hyponatremia remain clinically inconspicuous as the brain effectively adapts to the low extracellular osmolality. However, recent evidence suggests that even mild hyponatremia is associated with subtle neurocognitive deficits, gait disturbances, falls, fractures, and osteoporosis, as well as increased mortality. Current therapeutic interventions for hyponatremia, including fluid restriction and loop diuretics lack clinical trial data to support their efficacy and are commonly associated with poor adherence. The discovery of vasopressin antagonists (vaptans) provided a new drug class targeting the most common mechanism of hyponatremia, i.e., elevated vasopressin. Despite the demonstrated efficacy of vaptans in clinical trials, their use has been limited by high cost as well as safety concerns related to risk of liver injury and the potential for rapid correction of hyponatremia. Thus, despite the significant morbidity and mortality associated with chronic non-severe hyponatremia, there is a paucity of definitively effective, safe, well-tolerated, and reasonably priced treatments.

Small European case series have suggested that oral urea is safe and effective for the treatment of hyponatremia. However, urea has not been available for the treatment of hyponatremia in the United States until very recently. This research group recently published the first and only study describing the effectiveness and safety of a new American formulation of oral urea among hospitalized patients with hyponatremia. However, the latter was a retrospective study limited to hospitalized patients. Data from large clinical trials on the efficacy of urea for the prevention of patient-centered outcomes in those with chronic hyponatremia are lacking. The current proposal is a pilot study that seeks to establish the feasibility of recruiting ambulatory patients with chronic hyponatremia into a study of urea, determine the acceptability of urea to patients, and explore the effect of this agent on plasma sodium level (PNa), neurocognitive function, and postural stability. The investigators will recruit 30 ambulatory patients with chronic non-severe hyponatremia and randomize them to oral urea or no drug treatment for a period of 42 days. Following this initial phase, all participants will have a 10-day washout period, followed by a 42-day period in which participants initially randomized to no drug therapy will receive urea and those initially treated with urea will receive no drug therapy. The investigators will collect data regarding the ease of recruitment, participant adherence to urea, and adverse events related to its use. The investigators will monitor participants' PNa, neurocognitive function, and postural stability over the course of the study. The feasibility, acceptability, and proof of concept/efficacy data from this pilot study will confirm the investigator's capacity to conduct, and will inform the design of a large clinical trial that will assess the efficacy of urea for the prevention of serious clinical outcomes of chronic non-severe hyponatremia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Attended ≥1 visit at a University of Pittsburgh Medical Center (UPMC) outpatient clinic within the prior 12 months
* Chronic hyponatremia with a history of ≥ 2 sequential plasma sodium concentration (PNa) between 125 mmol/L and 132 mmol/L performed ≥ 14 days apart within the last 12 months with most recent PNa ≤ 132 mmol/L prior to screening
* Patients are ambulatory without the need for any assist device (e.g., cane, walker)
* Mini-mental state examination (MMSE) score ≥ 25
* Diagnosis of SIADH established by the Bartter and Schwartz criteria as follows:

  1. Hyponatremia with a PNa between 125 mmol/L and 132 mmol/L
  2. Plasma osmolality < 275 mOsm/kg
  3. Clinical euvolemia
  4. Urine osmolality > 100 mosm/kg
  5. Urine Na ≥ 20 mmol/L
  6. Intact adrenal function (i.e., morning plasma cortisol value ≥15 μg/dL, or negative corticotropin stimulation test)
  7. Normal thyroid stimulating hormone (TSH) level (i.e., TSH between 0.3 to 5 μIU/mL)
  8. eGFR >= 45 ml/min/1.73 m2)

Exclusion Criteria:

* Cirrhosis and/or end-stage liver disease
* Heart failure on diuretics and/or with recorded left ventricular ejection fraction <40 percent
* Chronic kidney disease with most recent estimated glomerular filtration rate <45 ml/min/1.73m2
* Adrenal insufficiency
* Untreated hypothyroidism
* Urinary tract obstruction within the prior 2 months
* Uncontrolled hyperglycemia (most recent random plasma glucose ≥ 200 mg/dL)
* Ongoing drug treatment for hyponatremia with vaptans or combination of loop diuretics and salt tablets.
* Active malignancy
* Active infection
* Neurological disorders with impairment of ambulation or cognition
* End-stage lung disease with marked impairment in ambulatory capacity
* Chronic pain with impairment of ambulation or cognition
* Chronic nausea
* Hypersensitivity to urea
* Women who are pregnant, breast feeding, or of childbearing potential who are not using contraception
* Patient is unable to consent for himself/herself

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helbert Rondon Berrios, MD. MS, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share all collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 12 months after publication of primary manuscript
Access Criteria: Request in writing addressed to the principal investigator

REFERENCES:
- [Background] Rondon-Berrios H, Berl T. Mild Chronic Hyponatremia in the Ambulatory Setting: Significance and Management. Clin J Am Soc Nephrol. 2015 Dec 7;10(12):2268-78. doi: 10.2215/CJN.00170115. Epub 2015 Jun 24. PMID 26109207
- [Background] Schrier RW, Gross P, Gheorghiade M, Berl T, Verbalis JG, Czerwiec FS, Orlandi C; SALT Investigators. Tolvaptan, a selective oral vasopressin V2-receptor antagonist, for hyponatremia. N Engl J Med. 2006 Nov 16;355(20):2099-112. doi: 10.1056/NEJMoa065181. Epub 2006 Nov 14. PMID 17105757
- [Background] Decaux G, Genette F. Urea for long-term treatment of syndrome of inappropriate secretion of antidiuretic hormone. Br Med J (Clin Res Ed). 1981 Oct 24;283(6299):1081-3. doi: 10.1136/bmj.283.6299.1081. PMID 6794768
- [Background] Rondon-Berrios H, Tandukar S, Mor MK, Ray EC, Bender FH, Kleyman TR, Weisbord SD. Urea for the Treatment of Hyponatremia. Clin J Am Soc Nephrol. 2018 Nov 7;13(11):1627-1632. doi: 10.2215/CJN.04020318. Epub 2018 Sep 4. PMID 30181129
- [Background] Gankam-Kengne F, Ayers C, Khera A, de Lemos J, Maalouf NM. Mild hyponatremia is associated with an increased risk of death in an ambulatory setting. Kidney Int. 2013 Apr;83(4):700-6. doi: 10.1038/ki.2012.459. Epub 2013 Jan 16. PMID 23325088
- [Background] Boscoe A, Paramore C, Verbalis JG. Cost of illness of hyponatremia in the United States. Cost Eff Resour Alloc. 2006 May 31;4:10. doi: 10.1186/1478-7547-4-10. PMID 16737547
- [Background] Decaux G. Is asymptomatic hyponatremia really asymptomatic? Am J Med. 2006 Jul;119(7 Suppl 1):S79-82. doi: 10.1016/j.amjmed.2006.05.013. PMID 16843090
- [Background] Renneboog B, Musch W, Vandemergel X, Manto MU, Decaux G. Mild chronic hyponatremia is associated with falls, unsteadiness, and attention deficits. Am J Med. 2006 Jan;119(1):71.e1-8. doi: 10.1016/j.amjmed.2005.09.026. PMID 16431193
- [Background] Verbalis JG, Barsony J, Sugimura Y, Tian Y, Adams DJ, Carter EA, Resnick HE. Hyponatremia-induced osteoporosis. J Bone Miner Res. 2010 Mar;25(3):554-63. doi: 10.1359/jbmr.090827. PMID 19751154
- [Background] Kruse C, Eiken P, Vestergaard P. Hyponatremia and osteoporosis: insights from the Danish National Patient Registry. Osteoporos Int. 2015 Mar;26(3):1005-16. doi: 10.1007/s00198-014-2973-1. Epub 2014 Dec 3. PMID 25466529
- [Background] Jamal SA, Arampatzis S, Harrison SL, Bucur RC, Ensrud K, Orwoll ES, Bauer DC. Hyponatremia and Fractures: Findings From the MrOS Study. J Bone Miner Res. 2015 Jun;30(6):970-5. doi: 10.1002/jbmr.2383. PMID 25294595
- [Background] Hoorn EJ, Rivadeneira F, van Meurs JB, Ziere G, Stricker BH, Hofman A, Pols HA, Zietse R, Uitterlinden AG, Zillikens MC. Mild hyponatremia as a risk factor for fractures: the Rotterdam Study. J Bone Miner Res. 2011 Aug;26(8):1822-8. doi: 10.1002/jbmr.380. PMID 21381111
- [Background] Mohan S, Gu S, Parikh A, Radhakrishnan J. Prevalence of hyponatremia and association with mortality: results from NHANES. Am J Med. 2013 Dec;126(12):1127-37.e1. doi: 10.1016/j.amjmed.2013.07.021. PMID 24262726
- [Background] Greenberg A, Verbalis JG, Amin AN, Burst VR, Chiodo JA 3rd, Chiong JR, Dasta JF, Friend KE, Hauptman PJ, Peri A, Sigal SH. Current treatment practice and outcomes. Report of the hyponatremia registry. Kidney Int. 2015 Jul;88(1):167-77. doi: 10.1038/ki.2015.4. Epub 2015 Feb 11. PMID 25671764
- [Background] Decaux G, Gankam Kengne F, Couturier B, Musch W, Soupart A, Vandergheynst F. Mild water restriction with or without urea for the longterm treatment of syndrome of inappropriate antidiuretic hormone secretion (SIADH): Can urine osmolality help the choice? Eur J Intern Med. 2018 Feb;48:89-93. doi: 10.1016/j.ejim.2017.09.024. Epub 2017 Oct 7. PMID 29017746
- [Background] Decaux G. Treatment of the syndrome of inappropriate secretion of antidiuretic hormone by long loop diuretics. Nephron. 1983;35(2):82-8. doi: 10.1159/000183052. No abstract available. PMID 6621759
- [Background] Decaux G, Waterlot Y, Genette F, Hallemans R, Demanet JC. Inappropriate secretion of antidiuretic hormone treated with frusemide. Br Med J (Clin Res Ed). 1982 Jul 10;285(6335):89-90. doi: 10.1136/bmj.285.6335.89. PMID 6805839
- [Background] Decaux G, Waterlot Y, Genette F, Mockel J. Treatment of the syndrome of inappropriate secretion of antidiuretic hormone with furosemide. N Engl J Med. 1981 Feb 5;304(6):329-30. doi: 10.1056/NEJM198102053040605. No abstract available. PMID 7442772
- [Background] Bhandari S, Peri A, Cranston I, McCool R, Shaw A, Glanville J, Petrakova L, O'Reilly K. A systematic review of known interventions for the treatment of chronic nonhypovolaemic hypotonic hyponatraemia and a meta-analysis of the vaptans. Clin Endocrinol (Oxf). 2017 Jun;86(6):761-771. doi: 10.1111/cen.13315. Epub 2017 Mar 27. PMID 28214374
- [Background] Jaber BL, Almarzouqi L, Borgi L, Seabra VF, Balk EM, Madias NE. Short-term efficacy and safety of vasopressin receptor antagonists for treatment of hyponatremia. Am J Med. 2011 Oct;124(10):977.e1-9. doi: 10.1016/j.amjmed.2011.04.028. PMID 21962320
- [Background] Li B, Fang D, Qian C, Feng H, Wang Y. The Efficacy and Safety of Tolvaptan in Patients with Hyponatremia: A Meta-Analysis of Randomized Controlled Trials. Clin Drug Investig. 2017 Apr;37(4):327-342. doi: 10.1007/s40261-016-0470-3. PMID 27766511
- [Background] Rozen-Zvi B, Yahav D, Gheorghiade M, Korzets A, Leibovici L, Gafter U. Vasopressin receptor antagonists for the treatment of hyponatremia: systematic review and meta-analysis. Am J Kidney Dis. 2010 Aug;56(2):325-37. doi: 10.1053/j.ajkd.2010.01.013. Epub 2010 Jun 9. PMID 20538391
- [Background] Zhang X, Zhao M, Du W, Zu D, Sun Y, Xiang R, Yang J. Efficacy and Safety of Vasopressin Receptor Antagonists for Euvolemic or Hypervolemic Hyponatremia: A Meta-Analysis. Medicine (Baltimore). 2016 Apr;95(15):e3310. doi: 10.1097/MD.0000000000003310. PMID 27082573
- [Background] Torres VE, Chapman AB, Devuyst O, Gansevoort RT, Grantham JJ, Higashihara E, Perrone RD, Krasa HB, Ouyang J, Czerwiec FS; TEMPO 3:4 Trial Investigators. Tolvaptan in patients with autosomal dominant polycystic kidney disease. N Engl J Med. 2012 Dec 20;367(25):2407-18. doi: 10.1056/NEJMoa1205511. Epub 2012 Nov 3. PMID 23121377
- [Background] Spasovski G, Vanholder R, Allolio B, Annane D, Ball S, Bichet D, Decaux G, Fenske W, Hoorn EJ, Ichai C, Joannidis M, Soupart A, Zietse R, Haller M, van der Veer S, Van Biesen W, Nagler E; Hyponatraemia Guideline Development Group. Clinical practice guideline on diagnosis and treatment of hyponatraemia. Nephrol Dial Transplant. 2014 Apr;29 Suppl 2:i1-i39. doi: 10.1093/ndt/gfu040. Epub 2014 Feb 25. PMID 24569496
- [Background] Decaux G, Andres C, Gankam Kengne F, Soupart A. Treatment of euvolemic hyponatremia in the intensive care unit by urea. Crit Care. 2010;14(5):R184. doi: 10.1186/cc9292. Epub 2010 Oct 14. PMID 20946646
- [Background] Lockett J, Berkman KE, Dimeski G, Russell AW, Inder WJ. Urea treatment in fluid restriction-refractory hyponatraemia. Clin Endocrinol (Oxf). 2019 Apr;90(4):630-636. doi: 10.1111/cen.13930. Epub 2019 Jan 25. PMID 30614552
- [Background] Nervo A, D'Angelo V, Rosso D, Castellana E, Cattel F, Arvat E, Grossi E. Urea in cancer patients with chronic SIAD-induced hyponatremia: Old drug, new evidence. Clin Endocrinol (Oxf). 2019 Jun;90(6):842-848. doi: 10.1111/cen.13966. Epub 2019 Mar 29. PMID 30868608
- [Background] Soupart A, Coffernils M, Couturier B, Gankam-Kengne F, Decaux G. Efficacy and tolerance of urea compared with vaptans for long-term treatment of patients with SIADH. Clin J Am Soc Nephrol. 2012 May;7(5):742-7. doi: 10.2215/CJN.06990711. Epub 2012 Mar 8. PMID 22403276
- [Background] Corona G, Giuliani C, Verbalis JG, Forti G, Maggi M, Peri A. Hyponatremia improvement is associated with a reduced risk of mortality: evidence from a meta-analysis. PLoS One. 2015 Apr 23;10(4):e0124105. doi: 10.1371/journal.pone.0124105. eCollection 2015. PMID 25905459
- [Background] Vandergheynst F, Gombeir Y, Bellante F, Perrotta G, Remiche G, Melot C, Mavroudakis N, Decaux G. Impact of hyponatremia on nerve conduction and muscle strength. Eur J Clin Invest. 2016 Apr;46(4):328-33. doi: 10.1111/eci.12597. Epub 2016 Feb 23. PMID 26835607
- [Background] Refardt J, Kling B, Krausert K, Fassnacht M, von Felten S, Christ-Crain M, Fenske W. Impact of chronic hyponatremia on neurocognitive and neuromuscular function. Eur J Clin Invest. 2018 Nov;48(11):e13022. doi: 10.1111/eci.13022. Epub 2018 Sep 19. PMID 30153330
- [Background] Verbalis JG, Greenberg A, Burst V, Haymann JP, Johannsson G, Peri A, Poch E, Chiodo JA 3rd, Dave J. Diagnosing and Treating the Syndrome of Inappropriate Antidiuretic Hormone Secretion. Am J Med. 2016 May;129(5):537.e9-537.e23. doi: 10.1016/j.amjmed.2015.11.005. Epub 2015 Nov 14. PMID 26584969
- [Background] Connaboy C, Johnson CD, LaGoy AD, Pepping GJ, Simpson RJ, Deng Z, Ma L, Bower JL, Eagle SR, Flanagan SD, Alfano CA. Intersession Reliability and Within-Session Stability of a Novel Perception-Action Coupling Task. Aerosp Med Hum Perform. 2019 Feb 1;90(2):77-83. doi: 10.3357/AMHP.5190.2019. PMID 30670116
- [Background] Erickson GB, Citek K, Cove M, Wilczek J, Linster C, Bjarnason B, Langemo N. Reliability of a computer-based system for measuring visual performance skills. Optometry. 2011 Sep;82(9):528-42. doi: 10.1016/j.optm.2011.01.012. Epub 2011 Jun 25. PMID 21705283
- [Background] Wang L, Krasich K, Bel-Bahar T, Hughes L, Mitroff SR, Appelbaum LG. Mapping the structure of perceptual and visual-motor abilities in healthy young adults. Acta Psychol (Amst). 2015 May;157:74-84. doi: 10.1016/j.actpsy.2015.02.005. Epub 2015 Mar 5. PMID 25747573
- [Background] Borg FG, Laxaback G. Entropy of balance--some recent results. J Neuroeng Rehabil. 2010 Jul 30;7:38. doi: 10.1186/1743-0003-7-38. PMID 20670457
- [Background] Kang HG, Costa MD, Priplata AA, Starobinets OV, Goldberger AL, Peng CK, Kiely DK, Cupples LA, Lipsitz LA. Frailty and the degradation of complex balance dynamics during a dual-task protocol. J Gerontol A Biol Sci Med Sci. 2009 Dec;64(12):1304-11. doi: 10.1093/gerona/glp113. Epub 2009 Aug 13. PMID 19679739
- [Background] Vereeck L, Wuyts F, Truijen S, Van de Heyning P. Clinical assessment of balance: normative data, and gender and age effects. Int J Audiol. 2008 Feb;47(2):67-75. doi: 10.1080/14992020701689688. PMID 18236239
- [Background] Wallmann HW. Comparison of elderly nonfallers and fallers on performance measures of functional reach, sensory organization, and limits of stability. J Gerontol A Biol Sci Med Sci. 2001 Sep;56(9):M580-3. doi: 10.1093/gerona/56.9.m580. PMID 11524452
- [Background] Sterns RH, Silver SM, Hix JK. Urea for hyponatremia? Kidney Int. 2015 Feb;87(2):268-70. doi: 10.1038/ki.2014.320. PMID 25635717
- See also: FDA Drug Safety Communication: FDA limits duration and usage of Samsca (tolvaptan) due to possible liver injury leading to organ transplant or death — https://www.fda.gov/drugs/drug-safety-and-availability/fda-drug-safety-communication-fda-limits-duration-and-usage-samsca-tolvaptan-due-possible-liver

RESULTS

PARTICIPANT FLOW:
Period: Period 1
Arm/Group | On Urea, Then Off Urea | Off Urea, Then On Urea
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0
Period: Washout Period
Arm/Group | On Urea, Then Off Urea | Off Urea, Then On Urea
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0
Period: Period 2
Arm/Group | On Urea, Then Off Urea | Off Urea, Then On Urea
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | On Urea, Then Off Urea | Off Urea, Then On Urea | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2
Plasma sodium concentration [Mean (Standard Deviation); unit: mmol/L] | 129 (NA) — 1 participant in each arm | 126 (NA) — 1 participant in each arm | 127.5 (2.1)
Accuracy action boundary selection [Mean (Standard Deviation); unit: percentage of accuracy] — Accuracy of affordance perception. Scores goes from 0% to 100% with higher score representing increased accuracy
  percentage of accuracy | 32.18 (NA) — Only 1 participant in each arm | 3.45 (NA) — Only 1 participant in each arm | 17.82 (20.3)
Score of sensorimotor ability battery [Mean (Standard Deviation); unit: units on a scale] — The Senaptec™ Sensory test battery was included to, in part, act as an azimuth check (i.e NFQ, CS, Visual Acuity, Depth Perception), for any changes in vision status cross the testing period, as this can influence balance control and potential fall risk. Additionally, some of the assessments provide insight into underlying sensorimotor process common to our active engagement with our surrounding environment (Reaction Time, MOT, Perception Span). Score goes from 0 to1500 with higher scores representing better sensorimotor ability
  units on a scale | 99.78 (NA) — Only 1 participant in each arm | 23.45 (NA) — Only 1 participant in each arm | 61.62 (54)
Sample entropy of the center of pressure data from the force plate [Mean (Standard Deviation); unit: percentage] — Measure the 'structure' of the noise in the oscillations of the center of mass of the individual. The measurement represent the percentage of displacement from the center of pressure. No reference ranges are available as these vary according to the population studied
  percentage | 6.7 (NA) — Only 1 participant in each arm | 0.2 (NA) — Only 1 participant in each arm | 3.45 (6)
Percentage angular deviation of vestibular control system using dynamic representation of upright st [Mean (Standard Deviation); unit: percentage] — The SOT consists of 6 conditions, each comprised of 3 trials lasting 20 sec each. Scores range between -100% to +200%. Lower percentage indicate poorer balance control
  percentage | 141.57 (NA) — Only 1 participant in each arm | 55.91 (NA) — Only 1 participant in each arm | 98.74 (61)
Percentage angular deviation of somatosensory control system using dynamic representation of upright [Mean (Standard Deviation); unit: percentage] — The SOT consists of 6 conditions, each comprised of 3 trials lasting 20 sec each. Scores range between -100% to +200%. Lower percentage indicate poorer balance control
  percentage | 0.05 (NA) — Only 1 participant in each arm | 2.11 (NA) — Only 1 participant in each arm | 1.08 (1)
Percentage angular deviation of visual control system using dynamic representation of upright stance [Mean (Standard Deviation); unit: percentage] — The SOT consists of 6 conditions, each comprised of 3 trials lasting 20 sec each. Scores range between -100% to +200%. Lower percentage indicate poorer balance control
  percentage | -2.53 (NA) — Only 1 participant in each arm | -5.9 (NA) — Only 1 participant in each arm | -4.22 (2)
Percentage weight symmetry using dynamic representation of upright stance [Mean (Standard Deviation); unit: percentage] — Weight symmetry indicates weight distribution under the left and right legs prior to perturbation onset. A score of 100 indicates perfect between-limb symmetry. Larger deviations away (higher or Lower) from 100 indicate asymmetry. Scores goes from -100% to +100% closer to 100% is optimal.
  percentage | -9.49 (NA) — Only 1 participant in each arm | 14.47 (NA) — Only 1 participant in each arm | 2.49 (17)
Movement latency of posture control and stability using dynamic representation of upright stance [Mean (Standard Deviation); unit: msec] — Latency scores measure the time lapse between force plate translation on postural response for healthy, elderly populations, with previously reported mean latency values ranging from 126.80-131.40. Higher/Larger scores indicate poorer balance control.
  msec | 4.598 (NA) — Only 1 participant in each arm | 8.331 (NA) — Only 1 participant in each arm | 6.46 (3)
Amplitude scaling of posture control and stability using dynamic representation of upright stance [Mean (Standard Deviation); unit: units on a scale] — The participant's ability to generate a response that is in proportion to the perturbation. It is scored in units of angular momentum and normalized to body height and weight. Scores range from 0 to 50 with values beyond a range of 0-15 are consider outside optimal
  units on a scale | 15.922 (NA) — Only 1 participant in each arm | 24.539 (NA) — Only 1 participant in each arm | 20.23 (6)
SF-12 (Health Survey) Mental Component Summary (MCS) [Mean (Standard Deviation); unit: units on a scale] — Scores range from 0 to 100, with higher scores indicating better mental health functioning
  units on a scale | 59.77660 (NA) — Only 1 participant in each arm | 57.92257 (NA) — Only 1 participant in each arm | 58.85 (1)
SF-12 (Health Survey) Physical Component Summary (PCS) [Mean (Standard Deviation); unit: units on a scale] — Scores range from 0 to 100, with higher scores indicating better physical health functioning
  units on a scale | 54.83583 (NA) — Only 1 participant in each arm | 53.79573 (NA) — Only 1 participant in each arm | 54.32 (1)

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Participants Who Met Inclusion/Exclusion Criteria and Were Enrolled in the Study
Description: Number and percentage of participants who met inclusion/exclusion criteria and were enrolled in the study. To be assessed by analysis of enrollment data.
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Groups:
- Urea; No Urea: Number and Percentage of Participants who Met Inclusion/Exclusion Criteria and were Enrolled in the Study
Arm/Group | Urea | No Urea
Number analyzed (Participants) | 2 | 2
Participants | 2 | 2

2. Primary Outcome: Number and Percentage of Participants Enrolled Who Completed the Study
Description: Number and percentage of participants enrolled who completed the study. To be assessed by analysis of enrollment and completion data.
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Groups:
- Urea; No Urea: Number and percentage of participants enrolled who completed the study.
Arm/Group | Urea | No Urea
Number analyzed (Participants) | 2 | 2
Participants | 2 | 2

3. Primary Outcome: Monthly Enrollment Rate
Description: Number of participants enrolled in the study every month. To be assessed by analysis of enrollment data
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: participants per month
Groups:
- Urea; No Urea: Monthly Enrollment Rate
Arm/Group | Urea | No Urea
Number analyzed (Participants) | 2 | 2
participants per month | 0.07 (0) | 0.07 (0)

4. Primary Outcome: Number of Prescribed Urea Doses Taken by Participants
Description: Number of prescribed urea doses taken by participants. To be assessed by records in study diary and number of returned medication doses.
Time Frame: Baseline to day 42 while taking urea
Population: The measure is only applicable when on urea
Measure: Mean (Full Range); unit: 15-g urea packets
Groups:
- Urea: Participants assigned to this group will receive oral urea for 42 days
Arm/Group | Urea
Number analyzed (Participants) | 2
15-g urea packets | 61.5 [11 to 112]

5. Primary Outcome: Reasons for Non-Adherence to Urea Therapy
Description: Reasons for non-adherence to urea therapy. To be assessed by medication acceptability and medication side effect questionnaires
Time Frame: Baseline to day 42 while taking urea
Population: The measure is only applicable when on urea
Measure: Count of Participants; unit: Participants
Arm/Group | Urea
Number analyzed (Participants) | 2
Participants
  Inconvenient medication dose frequency | 2
  Inconvenient medication amount | 1
  Medication is unsuitable to take outside home | 2
  Medication tastes poorly | 2
  Medications makes me feel sick | 1

6. Primary Outcome: Change in Plasma Sodium Concentration
Description: Change in plasma sodium concentration from baseline to day 42. Based on plasma sodium assessments on days 0 and 42.
Time Frame: Baseline to day 42
Population: All participants who received at least one dose of each intervention and completed all study visits were included
Measure: Mean (Full Range); unit: mmol/L
Groups:
- No Urea: Participants assigned to this group will be off urea for 42 days
Arm/Group | Urea | No Urea
Number analyzed (Participants) | 2 | 2
mmol/L | 2.5 [0 to 5] | 0.5 [0 to 1]

7. Primary Outcome: Change in Percentage Accuracy Action Boundary Selection
Description: Change in percentage accuracy action boundary selection from baseline to day 42. This will be measured by the Perception-Action Coupling Task (PACT) which is an affordance-based assessment conducted on an iPad, which uses matched pairs of 'virtual' balls and 'virtual' holes to assess patients' ability to accurately assess their action boundaries. Accuracy of affordance perception is measured. Scores goes from 0% to 100% with higher score representing increased accuracy
Time Frame: Baseline to day 42
Population: All participants who received at least one dose of each intervention and completed all study visits were included
Measure: Mean (Full Range); unit: percentage accuracy
Groups:
- No Urea: Participants assigned to this group will be off urea during for 42 days
Arm/Group | Urea | No Urea
Number analyzed (Participants) | 2 | 2
percentage accuracy | 12.965 [-6.25 to 32.18] | 8.245 [3.45 to 13.04]

8. Primary Outcome: Change in Overall Score of Sensorimotor Ability Battery
Description: Change in overall score of sensorimotor ability battery from baseline to day 42. This will be measured by the Senaptec Sensory Station™ test battery which examines separate sensorimotor elements including; multiple object tracking, reaction time, perception span, go/no go, depth perception and dynamic visual acuity. Score goes from 0 to1500 with higher scores representing better sensorimotor ability
Time Frame: Baseline to day 42
Population: All participants who received at least one dose of each intervention and completed all study visits were included
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Urea | No Urea
Number analyzed (Participants) | 2 | 2
score on a scale | 54.43 [9.09 to 99.78] | 53.6 [23.45 to 60.37]

9. Primary Outcome: Change in the Sample Entropy of the Center of Pressure Data From the Force Plate
Description: Measure the 'structure' of the noise in the oscillations of the center of mass of the individual. The measurement represent the percentage of displacement from the center of pressure. No reference ranges are available as these vary according to the population studied
Time Frame: Baseline to day 42
Population: All participants who received at least one dose of each intervention and completed all study visits were included
Measure: Mean (Full Range); unit: percentage change from baseline
Arm/Group | Urea | No Urea
Number analyzed (Participants) | 2 | 2
percentage change from baseline | 4.3 [1.9 to 6.7] | 1.3 [0.2 to 2.4]

10. Primary Outcome: Change in Percentage Angular Deviation of Vestibular Control System Using Dynamic Representation of Upright Stance
Description: Change in percentage angular deviation of vestibular control system using dynamic representation of upright stance from baseline to day 42. This was assessed using the NeuroCom™ Sensory Organization. This test enables both the examination of postural control and stability in response to a direct perturbation of the vestibular control system underlying the maintenance of upright posture, giving insight into the relative contributions and/or any deficits in the vestibular system involved in maintaining upright stance in dynamic situations. No reference range for changes in percentage exist which vary with the population studied. Larger positive changes indicate significant improvement in vestibular balance control.
Time Frame: Baseline to day 42
Population: All participants who received at least one dose of each intervention and completed all study visits were included
Measure: Mean (Full Range); unit: percentage
Arm/Group | Urea | No Urea
Number analyzed (Participants) | 2 | 2
percentage | 112.23 [82.9 to 141.57] | 88.0455 [55.91 to 120.19]

11. Primary Outcome: Change in Percentage Angular Deviation of Somatosensory Control System Using Dynamic Representation of Upright Stance
Description: Change in percentage angular deviation of somatosensory control system using dynamic representation of upright stance from baseline to day 42. This will be assessed using the NeuroCom™ Sensory Organization. This test enables both the examination of postural control and stability in response to a direct perturbation of the somatosensory control system underlying the maintenance of upright posture, giving insight into the relative contributions and/or any deficits in the somatosensory system involved in maintaining upright stance in dynamic situations. No reference range for changes in percentage exist which vary with the population studied. Larger positive changes indicate significant improvement in somatosensory balance control.
Time Frame: Baseline to day 42
Measure: Mean (Full Range); unit: percentage change from baseline
Arm/Group | Urea | No Urea
Number analyzed (Participants) | 2 | 2
percentage change from baseline | 1.99 [0.05 to 3.93] | -0.85 [-2.96 to 2.11]

12. Primary Outcome: Change in Percentage Angular Deviation of Visual Control System Using Dynamic Representation of Upright Stance
Description: Change in percentage angular deviation of visual control system using dynamic representation of upright stance from baseline to day 42. This will be assessed using the NeuroCom™ Sensory Organization. This test enables both the examination of postural control and stability in response to a direct perturbation of the visual control system underlying the maintenance of upright posture, giving insight into the relative contributions and/or any deficits in the visual system involved in maintaining upright stance in dynamic situations. No reference range for changes in percentage exist which vary with the population studied. Larger positive changes indicate significant improvement in visual balance control.
Time Frame: Baseline to 42 days
Measure: Mean (Full Range); unit: percentage change from baseline
Arm/Group | Urea | No Urea
Number analyzed (Participants) | 2 | 2
percentage change from baseline | -1.1735 [-2.53 to 0.19] | -7.3825 [-8.86 to -5.90]

13. Primary Outcome: Change in Percentage Weight Symmetry Using Dynamic Representation of Upright Stance
Description: Change in percentage weight symmetry using dynamic representation of upright stance from baseline to day 42. This will be assessed using the Motor Control Test (MCT). MCT assesses the ability to quickly recover from an unexpected external translation. Weight symmetry indicates weight distribution under the left and right legs prior to perturbation onset. A score of 100 indicates perfect between-limb symmetry. Larger deviations away (higher or Lower) from 100 indicate asymmetry. Scores goes from -100 to +100 closer to 100 is optimal.
Time Frame: Baseline to day 42
Measure: Mean (Full Range); unit: percentage change from baseline
Arm/Group | Urea | No Urea
Number analyzed (Participants) | 2 | 2
percentage change from baseline | -1.6255 [-9.49 to 6.24] | 2.5 [-9.47 to 14.47]

14. Primary Outcome: Change in Movement Latency of Posture Control and Stability Using Dynamic Representation of Upright Stance
Description: Change in movement latency of posture control and stability using dynamic representation of upright stance from baseline to day 42. This will be assessed using the Motor Control Test (MCT). MCT assesses the ability to quickly recover from an unexpected external translation. Latency scores measure the time lapse between force plate translation on postural response for healthy, elderly populations, with previously reported mean latency values ranging from 126.80-131.40. Higher/Larger scores indicate poorer balance control.
Time Frame: Baseline to day 42
Measure: Mean (Full Range); unit: milliseconds
Groups:
- No Urea: Participants assigned to this group will be off urea during 42 days
Arm/Group | Urea | No Urea
Number analyzed (Participants) | 2 | 2
milliseconds | -3.8245 [-12.247 to 4.598] | 8.677 [8.331 to 9.023]

15. Primary Outcome: Change in Amplitude Scaling of Posture Control and Stability Using Dynamic Representation of Upright Stance
Description: Change in amplitude scaling of posture control and stability using dynamic representation of upright stance from baseline to day 42. This will be assessed using the Motor Control Test (MCT). MCT assesses the ability to quickly recover from an unexpected external translation. It is scored in units of angular momentum and normalized to body height and weight. No reference range for changes in percentage exist which vary with the population studied. Larger positive changes indicate significant improvement in ability to recover from an unexpected external translation reflecting better balance.
Time Frame: Baseline to day 42
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Urea | No Urea
Number analyzed (Participants) | 2 | 2
units on a scale | 5.414 [-5.094 to 15.922] | 9.0495 [-6.44 to 24.539]

16. Primary Outcome: Number and Proportion of Participants Enrolled in the Study With Adverse Events Related to the Use of Urea
Description: Number and proportion of participants enrolled in the study with adverse events related to the use of urea from baseline to day 42. To be assessed by medication side effect questionnaire.
Time Frame: Baseline to day 42 while taking urea
Population: This measure is only relevant when on urea
Measure: Count of Participants; unit: Participants
Arm/Group | Urea | No Urea
Number analyzed (Participants) | 2 | 2
Participants | 1 | 0

17. Primary Outcome: Adverse Events Related to Urea
Description: To be assessed by medication side effect questionnaire. A tabulation of counts of participants experiencing specific known side effects of urea as well as their intensity (mild, moderate or severe) will be performed.
Time Frame: Baseline to day 42 while taking urea
Population: The measure is only applicable when on urea
Measure: Count of Participants; unit: Participants
Groups:
- Urea: Participants received oral urea for 42 days
Arm/Group | Urea
Number analyzed (Participants) | 2
Participants
  Nausea: None | 1
  Nausea: Mild | 0
  Nausea: Moderate | 1
  Nausea: Severe | 0
  Vomiting: None | 2
  Vomiting: Mild | 0
  Vomiting: Moderate | 0
  Vomiting: Severe | 0
  Diarrhea: None | 1
  Diarrhea: Mild | 1
  Diarrhea: Moderate | 0
  Diarrhea: Severe | 0
  Headaches: None | 1
  Headaches: Mild | 0
  Headaches: Moderate | 1
  Headaches: Severe | 0

18. Secondary Outcome: Number of Patients Screened
Description: Number of patients screened. To be assessed by analysis of screening data.
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Groups:
- Number of Patients Screened: Number of patients screened.
Arm/Group | Number of Patients Screened
Number analyzed (Participants) | 1213
Participants | 1213

19. Secondary Outcome: Number and Percentage of Patients Screened Who Met Inclusion/Exclusion Criteria for the Study
Description: Number and percentage of patients screened who met inclusion/exclusion criteria for the study.
  To be assessed by analysis of screening and enrollment data.
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Groups:
- Number and Proportion of Patients Screened Who Met Inclusion/Exclusion Criteria for the Study: Number and proportion of patients screened who met inclusion/exclusion criteria for the study. To be assessed by analysis of screening data
Arm/Group | Number and Proportion of Patients Screened Who Met Inclusion/Exclusion Criteria for the Study
Number analyzed (Participants) | 1213
Participants | 2

20. Secondary Outcome: Number and Proportion of Participants Who Took More Than 80 Percent of Prescribed Urea Doses
Description: Number and proportion of participants who took more than 80 percent of prescribed urea doses. To be assessed by analysis of study diary and number of returned medication doses.
Time Frame: Baseline to day 42 while taking urea
Population: All participants who received at least one dose of each intervention and completed all study visits were included. The measure is only applicable when on urea.
Measure: Count of Participants; unit: Participants
Arm/Group | Urea
Number analyzed (Participants) | 2
Participants | 1

21. Secondary Outcome: Number and Proportion of Participants Who Thought the Medication Was Acceptable
Description: Number and proportion of participants who thought the medication was acceptable. Based on ratings for acceptability in the medication acceptability questionnaire.
Time Frame: Baseline to day 42 while taking urea
Population: All participants who received at least one dose of each intervention and completed all study visits were included
Measure: Count of Participants; unit: Participants
Arm/Group | Urea | No Urea
Number analyzed (Participants) | 2 | 2
Participants | 1 | 0

22. Secondary Outcome: Average Ratings for Medication Acceptability
Description: Average ratings using a 5-point Likert scale medication acceptability questionnaire. in which responders specify their level of agreement to a statement in five points: (1) Strongly disagree; (2) Disagree; (3) Neutral; (4) Agree; (5) Strongly agree; or (1) Very Unhappy; (2) Unhappy; (3) Neutral; (4) Happy; (5) Very Happy. A higher overall score represents more acceptability
Time Frame: Baseline to day 42 while taking urea
Population: The measure is only applicable when on urea
Measure: Mean (Full Range); unit: units on a 5-point Likert scale
Arm/Group | Urea
Number analyzed (Participants) | 2
units on a 5-point Likert scale | 2.725 [1 to 5]

23. Secondary Outcome: Change in SF-12 (Health Survey) Mental Component Summary (MCS)
Description: Change in SF-12 (Health Survey) Mental Component Summary (MCS) from baseline to day 42. Based on SF-12 MCS assessments on days 0 and 42. This is computed using the scores of 12 questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Time Frame: Baseline to day 42
Population: All participants who received at least one dose of each intervention and completed all study visits were included
Measure: Mean (Full Range); unit: score on SF-12 scale
Arm/Group | Urea | No Urea
Number analyzed (Participants) | 2 | 2
score on SF-12 scale | 1.435 [0.90384 to 1.95934] | 0.745 [0.59 to 0.90384]

24. Secondary Outcome: Change in SF-12 (Health Survey) Physical Component Summary (PCS)
Description: Change in SF-12 (Health Survey) Physical Component Summary (PCS) from baseline to day 42. Based on SF-12 PCS assessments on days 0 and 42. This is computed using the scores of 12 questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Time Frame: Baseline to day 42
Population: All participants who received at least one dose of each intervention and completed all study visits were included
Measure: Mean (Full Range); unit: score on a SF-12 scale
Arm/Group | Urea | No Urea
Number analyzed (Participants) | 2 | 2
score on a SF-12 scale | -2.105 [-3.8 to -0.41] | -3.25 [-3.8 to -2.7]

ADVERSE EVENTS:
Time Frame: 94 days
Arm/Group | Urea | No Urea
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Urea (N=2) | No Urea (N=2)
Nausea (Gastrointestinal disorders) | 1 (4) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headaches (Nervous system disorders) | 1 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (3) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was terminated because of inability to recruit. Only two participants were recruited of the estimated 30 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-25): https://cdn.clinicaltrials.gov/large-docs/07/NCT04588207/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/07/NCT04588207/ICF_001.pdf